CLINICAL TRIAL: NCT05693246
Title: Effect of Perioperative Use of Glycopyrrolate on Lung Function in Patients Under General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, :: Principal Investigator, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20221202
Record Dates: First submitted 2022-12-03; First posted 2023-01-20 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Glycopyrrolate
Keywords: Glycopyrrolate; Perioperative period; Lung compliance; Autonomic nervous system
MeSH Terms: interventions — Glycopyrrolate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glycopyrrolate (Experimental)
  Interventions: Drug: Glycopyrrolate
- Control (Placebo Comparator)
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: Glycopyrrolate — At 10 minutes after endotracheal intubation, the Glycopyrrolate group was injected intravenously with 0.004mg/kg glycopyrrolate.
  Arms: Glycopyrrolate
Other: normal saline — At 10 minutes after endotracheal intubation, the Control group was intravenously injected with equal dose of normal saline.
  Arms: Control

SUMMARY:
Gastrointestinal tumor is one of the highest incidence of malignant tumors in our country, with the incidence increasing year by year. Laparoscopic gastrointestinal surgery ,due to having less bleeding ,small trauma ,Rapid recovery ,has become the main means for the treatment of gastrointestinal surgery. Under general anesthesia, mechanical ventilation can lead to repeated mechanical dilation of alveoli, which can lead to mechanical injury of alveolar epithelium, reduce lung compliance, affect lung function, and increase postoperative complications and hospital stay of patients. Glycopyrrolate acts selectively on M1 and M3 receptors, and is 3-5 times more selective to M3 and M1 receptors than M2 receptors. Therefore, as preoperative medication for elderly patients, it has less effect on the cardiovascular system and can stabilize the heart rate,compared with atropine.However, its influence on the respiratory system in the field of anesthesia is only limited to the study of inhibiting glandular secretion at present, and there are no clear reports on the study of respiratory mechanics .The purpose of this study was to investigate the effects of glycopyrrolate on lung function and respiratory mechanics in elderly patients after general anesthesia, in order to guide clinical medication.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients undergoing elective laparoscopic radical surgery for gastrointestinal malignant tumors;
2. ASA Grade I-III;
3. BMI 18 to 30 kg /㎡；
4. Operation time≥2 hours.

Exclusion Criteria:

1. Hypersensitivity to glycopyrrolate；
2. Clinical diagnosis of hepatic and renal insufficiency；
3. Complicated myasthenia gravis；
4. Prolonged QT interval and other abnormal electrocardiogram；
5. History of mechanical ventilation within six months before surgery；
6. Combined with glaucoma；
7. The patient refused.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
the changes in lung compliance | 10 minutes after intubation; 10 minutes after pneumoperitoneum; 1 hour after pneumoperitoneum; End of pneumoperitoneum for 10 minutes
  Lung compliance refers to the degree to which the lungs change under external forces

SECONDARY OUTCOMES:
the changes in oxygenation index | 10 minutes after intubation; 10 minutes after pneumoperitoneum; 1 hour after pneumoperitoneum; End of pneumoperitoneum for 10 minutes
  Oxygenation index is an important indicator of lung function

OTHER OUTCOMES:
the changes in systolic blood pressure | 10 minutes after intubation;10 minutes after pneumoperitoneum; 1 hour after pneumoperitoneum; End of pneumoperitoneum for 10 minutes
  Record changes in systolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China